CLINICAL TRIAL: NCT02248324
Title: A Multicenter Study on the Investigation of Previously Verified Leading Gene Polymorphisms Related to Age-related Macular Degeneration in Turkish Population
Brief Title: Association of Previously Verified Gene Polymorphisms With AMD in Turkish Population
Acronym: AMD-SNP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocatepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Umit Ubeyt INAN, Professor Doctor, Kocatepe University
Other Study IDs: 0112S269
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related macular degeneration, genetic polymorphisms
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether common genetic polymorphisms that have been verified to be related to age-related macular degeneration (AMD) in some populations are also associated with AMD in Turkish population

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) remains as the most important cause of severe visual impairment of elderly people in developed countries. It is one of the best-characterized complex trait diseases. Multiple genetic and environmental factors play a role in the pathogenesis. A number of different biological pathways and related gene polymorphisms are strongly implicated in its etiology. A lot of chromosomal locations have been studied to figure out genetic risk factors responsible from the development of AMD. Most genetic variants that have been found to be related to AMD at least in one study have not been verified in subsequent studies. However in recent years, single-nucleotide polymorphisms related to the complement system and also chromosome 10q26 have strongly been elicited to predispose individuals to the susceptibility to AMD. These polymorphisms have been verified in subsequent studies. However, results from different geographic regions of the world can represent discrepancies according to ethnic populations. Aforementioned genetic tests have been commercially introduced to give the patients the risk of progression to advanced stage of AMD, and rate of the risk can be given by the genetic results together with environmental factors in USA.

Age related macular degeneration is consisted of dry and wet forms. Although wet form is responsible from severe vision loss due to AMD, dry form can progress to wet form by passage of time. The risk of AMD increases when age get older and it causes very severe central vision loss; consequently reduces considerably the quality of life in senile population. Available treatment of AMD is expensive and has economical burden. Early diagnosis of the disease has favourable impact on post-treatment prognosis. Although the basis of treatment is primarily based on the preservation of current visual acuity, it is possible to obtain improvement in visual acuity with the agents inhibiting angiogenesis in recent years. However, complete response to the treatment is not obtained approximately in one fifth of the patients. Different responses to the treatment are obtained in the remaining group. The reason for the differences at the treatment may be due to different morphological subgroups and/or diversity of genetic variants in wet AMD. . We do not at the moment know whether gen polymorphisms related to AMD established in some western population are also related to AMD in our population or whether this relationship has similar risk or protective effect for AMD. The gen variants mostly studied in relation to AMD are CFH (rs1061170 and rs1410996), LOC387715/ARMS-2 (A69S /rs10490924), HTRA-1 (rs11200638), C3 (R102G/ rs2230199), C2 E318D (rs9332739), and CFB R32Q (rs641153). A preliminary study which was published recently, carried out by our team in a single center and in a small number of patients showed that CFH and LOC387715 gen polymorphisms entertain a risk for late AMD and suggested a necessity to perform a forward study with larger population to learn definite information about our population. On the other hand, the entire eight genetic locus related to AMD will be studied first time in our population. In the introduced projects study, the relationship of eight different gen polymorphisms (CFH rs1061170 and rs1410996, LOC387715 / ARMS2 gene rs10490924, C2 gene rs9332739, CFB gene rs641153, CFI rs10033900 , HTRA-1 gene rs11200638, C3 rs2230199) will be studied in 2800 patients with high risk intermediate and late stage AMD and 2200 age-matched control subjects. Blood samples from brachial veins of the study subjects will be collected in the 5 health centers composed of Bursa Retina Eye Center and Hospitals of Afyon Kocatepe University, Dokuz Eylul University, Konya University and Uludag University within the period of 32 months. After the collection of venous samples, polymorphisms will be genotyped by "real-time PCR'' and ''pyrosequencing" genotyping systems in the genetic laboratory of Afyon Kocatepe University Medical School. Within the last 3 months of the project duration, having completed genotyping of all samples, evaluation of the study data by clinically and statistically will be made, and preparation of final report will be realized. . As a primary outcome, protective effects or the risk rate of developing the late AMD for each genetic polymorphism will be calculated by statistical analysis following the genotyping. Sub-analyses will be done to investigate any relationship between genetic polymorphism and response to the treatment. Sub-analyses will be done to determine possible differences in genetic variants between the late dry and wet AMD and also among the morphological subtypes of the wet AMD. Main study and secondary sub-studies derived from sub-analyses by further methodology will be submitted as different studies for publication. The anticipated results of the study may have impact on the management and follow-up of the patients with AMD. Because AMD is etiologically multi-factorial disease and has environmental controllable risk factor outside the genotypic features, it may be possible to early diagnosis and frequent follow-up in addition to recommending to avoid from modifiable risk factors in patients with early AMD who are genetically under the high risk of the development of late AMD according to findings obtained from our study results. It will also be possible to establish the patients with wet AMD who are resistant or sensitive to the treatment according to genotyping. Whether performing genetic tests in patients who are candidate to the late AMD in the near future is significant and meaningful for our population will be established. Our results evaluated together with the literature will make substantial contribution to better understanding of pathogenesis of AMD as well as early diagnosis and better classification or treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Older age more than 50 years for the study group and older age more than 60 years for the control group
* Intermediate or advanced stage age-related macular degeneration
* Active or inactive scar choroidal neovascularization
* For control patients: Normal macular anatomy and no sign of any stage of age-related macular degeneration

Exclusion Criteria:

* People with findings of advanced age-related macular degeneration due to other reasons (inflammatory, myopic choroidal neovascularization etc..)
* For control patients: Any sign of age-related macular degeneration

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate and advanced age related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
rate of homozygous, heterozygous or wild type genotype and allels | at the end of third years
  Gene polymorphisms of 8 region with identification of homozygous, heterozygote and wild type genotyping and alleles

SECONDARY OUTCOMES:
Odds ratios for each genotyping in healthy elderly controls and patients with age related macular degeneration | at the end of third years

OTHER OUTCOMES:
Odds ratios for various combinations of gene regions between healthy elderly control and patients with age related macular degeneration | at the end of third years

CONTACTS AND LOCATIONS:
Overall Officials: Umit U INAN, MD, Study Chair — Kocatepe University Medical School Department of Ophthalmology
Locations (1):
- Umit Ubeyt INAN, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Result] Kim YH, Kim HS, Mok JW, Joo CK. Gene-gene interactions of CFH and LOC387715/ARMS2 with Korean exudative age-related macular degeneration patients. Ophthalmic Genet. 2013 Sep;34(3):151-9. doi: 10.3109/13816810.2012.749287. Epub 2013 Jan 4. PMID 23289807
- [Result] Xu Y, Guan N, Xu J, Yang X, Ma K, Zhou H, Zhang F, Snellingen T, Jiao Y, Liu X, Wang N, Liu N. Association of CFH, LOC387715, and HTRA1 polymorphisms with exudative age-related macular degeneration in a northern Chinese population. Mol Vis. 2008 Jul 28;14:1373-81. PMID 18682812
- [Result] Francis PJ, Zhang H, Dewan A, Hoh J, Klein ML. Joint effects of polymorphisms in the HTRA1, LOC387715/ARMS2, and CFH genes on AMD in a Caucasian population. Mol Vis. 2008 Aug 4;14:1395-400. PMID 18682806
- [Result] Jakobsdottir J, Conley YP, Weeks DE, Ferrell RE, Gorin MB. C2 and CFB genes in age-related maculopathy and joint action with CFH and LOC387715 genes. PLoS One. 2008 May 21;3(5):e2199. doi: 10.1371/journal.pone.0002199. PMID 18493315
- [Result] Kaur I, Katta S, Hussain A, Hussain N, Mathai A, Narayanan R, Hussain A, Reddy RK, Majji AB, Das T, Chakrabarti S. Variants in the 10q26 gene cluster (LOC387715 and HTRA1) exhibit enhanced risk of age-related macular degeneration along with CFH in Indian patients. Invest Ophthalmol Vis Sci. 2008 May;49(5):1771-6. doi: 10.1167/iovs.07-0560. PMID 18436811
- [Result] Klein ML, Francis PJ, Rosner B, Reynolds R, Hamon SC, Schultz DW, Ott J, Seddon JM. CFH and LOC387715/ARMS2 genotypes and treatment with antioxidants and zinc for age-related macular degeneration. Ophthalmology. 2008 Jun;115(6):1019-25. doi: 10.1016/j.ophtha.2008.01.036. PMID 18423869
- [Result] Hughes AE, Orr N, Patterson C, Esfandiary H, Hogg R, McConnell V, Silvestri G, Chakravarthy U. Neovascular age-related macular degeneration risk based on CFH, LOC387715/HTRA1, and smoking. PLoS Med. 2007 Dec;4(12):e355. doi: 10.1371/journal.pmed.0040355. PMID 18162041
- [Result] Seddon JM, Francis PJ, George S, Schultz DW, Rosner B, Klein ML. Association of CFH Y402H and LOC387715 A69S with progression of age-related macular degeneration. JAMA. 2007 Apr 25;297(16):1793-800. doi: 10.1001/jama.297.16.1793. PMID 17456821
- [Result] Seddon JM, Reynolds R, Maller J, Fagerness JA, Daly MJ, Rosner B. Prediction model for prevalence and incidence of advanced age-related macular degeneration based on genetic, demographic, and environmental variables. Invest Ophthalmol Vis Sci. 2009 May;50(5):2044-53. doi: 10.1167/iovs.08-3064. Epub 2008 Dec 30. PMID 19117936
- [Result] Seddon JM, George S, Rosner B, Klein ML. CFH gene variant, Y402H, and smoking, body mass index, environmental associations with advanced age-related macular degeneration. Hum Hered. 2006;61(3):157-65. doi: 10.1159/000094141. Epub 2006 Jun 30. PMID 16816528
- [Result] Brantley MA Jr, Fang AM, King JM, Tewari A, Kymes SM, Shiels A. Association of complement factor H and LOC387715 genotypes with response of exudative age-related macular degeneration to intravitreal bevacizumab. Ophthalmology. 2007 Dec;114(12):2168-73. doi: 10.1016/j.ophtha.2007.09.008. PMID 18054635
- [Result] Despriet DD, van Duijn CM, Oostra BA, Uitterlinden AG, Hofman A, Wright AF, ten Brink JB, Bakker A, de Jong PT, Vingerling JR, Bergen AA, Klaver CC. Complement component C3 and risk of age-related macular degeneration. Ophthalmology. 2009 Mar;116(3):474-480.e2. doi: 10.1016/j.ophtha.2008.09.055. Epub 2009 Jan 24. PMID 19168221
- [Result] Francis PJ, George S, Schultz DW, Rosner B, Hamon S, Ott J, Weleber RG, Klein ML, Seddon JM. The LOC387715 gene, smoking, body mass index, environmental associations with advanced age-related macular degeneration. Hum Hered. 2007;63(3-4):212-8. doi: 10.1159/000100046. Epub 2007 Mar 7. PMID 17347568
- [Result] Seitsonen SP, Onkamo P, Peng G, Xiong M, Tommila PV, Ranta PH, Holopainen JM, Moilanen JA, Palosaari T, Kaarniranta K, Meri S, Immonen IR, Jarvela IE. Multifactor effects and evidence of potential interaction between complement factor H Y402H and LOC387715 A69S in age-related macular degeneration. PLoS One. 2008;3(12):e3833. doi: 10.1371/journal.pone.0003833. Epub 2008 Dec 2. PMID 19048105
- [Result] Francis PJ, Hamon SC, Ott J, Weleber RG, Klein ML. Polymorphisms in C2, CFB and C3 are associated with progression to advanced age related macular degeneration associated with visual loss. J Med Genet. 2009 May;46(5):300-7. doi: 10.1136/jmg.2008.062737. Epub 2008 Nov 17. PMID 19015224
- [Result] Caire J, Recalde S, Velazquez-Villoria A, Garcia-Garcia L, Reiter N, Anter J, Fernandez-Robredo P, Alfredo Garcia-Layana; Spanish Multicenter Group on AMD. Growth of geographic atrophy on fundus autofluorescence and polymorphisms of CFH, CFB, C3, FHR1-3, and ARMS2 in age-related macular degeneration. JAMA Ophthalmol. 2014 May;132(5):528-34. doi: 10.1001/jamaophthalmol.2013.8175. PMID 24557084
- [Result] Shuler RK Jr, Hauser MA, Caldwell J, Gallins P, Schmidt S, Scott WK, Agarwal A, Haines JL, Pericak-Vance MA, Postel EA. Neovascular age-related macular degeneration and its association with LOC387715 and complement factor H polymorphism. Arch Ophthalmol. 2007 Jan;125(1):63-7. doi: 10.1001/archopht.125.1.63. PMID 17210853
- [Result] Wegscheider BJ, Weger M, Renner W, Steinbrugger I, Marz W, Mossbock G, Temmel W, El-Shabrawi Y, Schmut O, Jahrbacher R, Haas A. Association of complement factor H Y402H gene polymorphism with different subtypes of exudative age-related macular degeneration. Ophthalmology. 2007 Apr;114(4):738-42. doi: 10.1016/j.ophtha.2006.07.048. PMID 17398321
- [Result] Seddon JM, Reynolds R, Yu Y, Daly MJ, Rosner B. Risk models for progression to advanced age-related macular degeneration using demographic, environmental, genetic, and ocular factors. Ophthalmology. 2011 Nov;118(11):2203-11. doi: 10.1016/j.ophtha.2011.04.029. Epub 2011 Sep 29. PMID 21959373
- [Result] Andreoli MT, Morrison MA, Kim BJ, Chen L, Adams SM, Miller JW, DeAngelis MM, Kim IK. Comprehensive analysis of complement factor H and LOC387715/ARMS2/HTRA1 variants with respect to phenotype in advanced age-related macular degeneration. Am J Ophthalmol. 2009 Dec;148(6):869-74. doi: 10.1016/j.ajo.2009.07.002. Epub 2009 Oct 1. PMID 19796758
- [Result] Sofat R, Casas JP, Webster AR, Bird AC, Mann SS, Yates JR, Moore AT, Sepp T, Cipriani V, Bunce C, Khan JC, Shahid H, Swaroop A, Abecasis G, Branham KE, Zareparsi S, Bergen AA, Klaver CC, Baas DC, Zhang K, Chen Y, Gibbs D, Weber BH, Keilhauer CN, Fritsche LG, Lotery A, Cree AJ, Griffiths HL, Bhattacharya SS, Chen LL, Jenkins SA, Peto T, Lathrop M, Leveillard T, Gorin MB, Weeks DE, Ortube MC, Ferrell RE, Jakobsdottir J, Conley YP, Rahu M, Seland JH, Soubrane G, Topouzis F, Vioque J, Tomazzoli L, Young I, Whittaker J, Chakravarthy U, de Jong PT, Smeeth L, Fletcher A, Hingorani AD. Complement factor H genetic variant and age-related macular degeneration: effect size, modifiers and relationship to disease subtype. Int J Epidemiol. 2012 Feb;41(1):250-62. doi: 10.1093/ije/dyr204. Epub 2012 Jan 13. PMID 22253316
- [Result] Klein R, Myers CE, Meuer SM, Gangnon RE, Sivakumaran TA, Iyengar SK, Lee KE, Klein BE. Risk alleles in CFH and ARMS2 and the long-term natural history of age-related macular degeneration: the Beaver Dam Eye Study. JAMA Ophthalmol. 2013 Mar;131(3):383-92. doi: 10.1001/jamaophthalmol.2013.713. PMID 23494043
- [Result] Lima LH, Schubert C, Ferrara DC, Merriam JE, Imamura Y, Freund KB, Spaide RF, Yannuzzi LA, Allikmets R. Three major loci involved in age-related macular degeneration are also associated with polypoidal choroidal vasculopathy. Ophthalmology. 2010 Aug;117(8):1567-70. doi: 10.1016/j.ophtha.2009.12.018. Epub 2010 Apr 8. PMID 20378180